CLINICAL TRIAL: NCT04425083
Title: Study of the Relationship of the Chinese Medical Constitution & Syndromes and Quality of Life in Patients With Polycystic Ovary Syndrome
Brief Title: Relationship of the Chinese Medical Constitution & Syndromes in Patients With Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chien-Jung Lin, department of Chinese medicine, Tri-Service General Hospital
Other Study IDs: TSGH-C105-025
Record Dates: First submitted 2020-05-23; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Chinese Medical Constitution & Syndromes
MeSH Terms: conditions — Polycystic Ovary Syndrome; Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polycystic Ovary Syndrome: Polycystic Ovary Syndrome women
  Interventions: Other: no intervention
- control: non- Polycystic Ovary Syndrome women
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study is a cross-sectional study. The purpose is to understand the characteristics of Chinese medicine constitutional syndrome in patients with polycystic ovary. In addition, the health-related quality of life (SF-36), mental state (stress, depression) of patients with polycystic ovary , Anxiety) and the relationship between hormone biochemical indicators and TCM constitutional syndromes, to develop a pioneering study on TCM constitution diagnosis and life guidelines for polycystic ovarian patients and future clinical adjuvant therapy.

DETAILED DESCRIPTION:
The study conducted in the Obstetrics and Gynecology Department of the Neihu District of the Taipei Three Military General Hospital. It is expected that 200 cases of polycystic ovary will be diagnosed by specialists; "Quality of Life Questionnaire (SF-36)" evaluates the quality of life of patients; "BAI and BDI-II" evaluates patients 'anxiety and depression; "Stress Perception Scale" evaluates patients' life stress And testing the blood indexes of patients such as FSH, LH, E2, testosterone, TSH, prolactine. Observe the correlation between the quality of life, psychological state, and blood test values of polycystic ovarian patients with physical characteristics of traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

A polycystic ovarian patient was diagnosed by a specialist in obstetrics and gynecology according to the diagnostic criteria set by the Rotterdam ESHRE / ASRM-sponsored PCOS workshop group (2004) in 2003.

Exclusion Criteria:

1. Exclude diseases similar to the clinical manifestations of polycystic ovary, such as cushing syndrome, congenital adrenal hyperplasia, thyroid dysfunction, and hyperprolactinemia.
2. Diagnose a clear mental disorder (such as schizophrenia, severe depression) or take psychiatric drugs (anti-depression or anxiety drugs).
3. Pregnancy, oral contraceptives, use high-dose exogenous androgens, breastfeeding.
4. Those with a history of stroke, myocardial infarction, major trauma or surgery within the past six months.
5. Have taken Chinese medicine in the past month.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with Polycystic Ovary Syndrome and non Polycystic Ovary Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
participants with PCOS and non-PCOS assessed Chinese Body Constitution & Syndromes by Body Constitution Questionnaire | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  The TCM Body Constitution Questionnaire (BCQ) was developed by Su and is a tool used to measure and study constitution deviations clinically. The questionnaire comprises 44 questions and employs a Likert 5-point scale (from 1, "Never happens," to 5, "Always happens"). The instrument consists of three subscales. The yang-xu and yin-xu constitution subscales each have 19 questions, and the stasis constitution subscale has 16 questions. The three measures share some questions. The higher the score is, the more significant the constitution deviation is. When the yang-xu constitution score is ≥ 30.5, the respondent is diagnosed as yang-xu. When the yin-xu constitution score is ≥ 29.5, the respondent is diagnosed as yin-xu. For the phlegm stasis constitution, the standard is ≥ 26.5 points. The instrument has favorable factorial validity. Cronbach's α of each subscale is 0.85-0.88, and Cronbach's αof the overall BCQ reaches 0.90.

SECONDARY OUTCOMES:
work schedule (Day shift, Evening shift, Night shift, Not fixed, or Unemployed) of participants with PCOS and non-PCOS were collected | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  Participant reply her work schedule (Day shift, Evening shift, Night shift, Not fixed, or Unemployed)
average sleep duration of participants with PCOS and non-PCOS were collected | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  Participant reply her average sleep duration (hours)
habit of staying up late of participants with PCOS and non-PCOS were collected | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  Participant reply her frequency(No, Sometimes, Often) of staying up late (sleeping after midnight)
habit of smoking of participants with PCOS and non-PCOS were collected | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  Participant reply her frequency of smoking (No, Sometimes, Less than a pack a day)
habit of drinking of participants with PCOS and non-PCOS were collected | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  Participant reply her frequency of drinking (No, Sometimes, often)
habit of exercise of participants with PCOS and non-PCOS were collected | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  Participant reply her frequency of exercise (No, Sometimes, often)
dietary habit (Nonvegetarian or vegetarian) of participants with PCOS and non-PCOS were collected | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  Participant reply her dietary habit (Nonvegetarian or vegetarian)
dietary flavor preference (sour, bitter,sweet, spicy, salty) of participants with PCOS and non-PCOS were collected | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  Participant reply yes or no about her dietary flavor preference (sour, bitter,sweet, spicy, salty)
Anxiety of participants with PCOS and non-PCOS as assessed by Beck Anxiety Inventory | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  The Beck Anxiety Inventory (BAI) was established by Aaron T. Beck and his research team to measure the anxiety levels of adults and teenagers. It is a self-completed questionnaire with 21 items. The questions ask respondents whether they have experienced some common symptoms of anxiety in the previous week, including numbness or tingling, feeling hot, being unable to relax, and fear of the worst happening. The respondents report on a 4-point Likert scale that ranges from 0 (Not at all) to 3 (Severely - it bothered me a lot). The higher the total score is, the more severe the anxiety symptoms are. A total score of 0-7 implies the mildest anxiety, 8-15 is mild anxiety, 16-25 represents moderate anxiety, and 26-63 is severe anxiety. In the present study, the Chinese version of the BAI had a Cronbach's α of 0.95 and a split-half reliability of 0.92. The total scores were multiplied by 1.19, and the resulted integers were taken as the standard scores.
Depression of participants with PCOS and non-PCOS as assessed by Beck Depression Inventory-second edition (BDI-II) | No subsequent intervention, data collected and analyzed at the time of enrolled (cross-sectional study)
  The Beck Depression Inventory-second edition (BDI-II) was developed by Beck . It measures the depression levels of teenagers and adults through 21 questions. It consists of questions representative of the symptoms and attitudes of depression, such as feeling sad, losing interest, decreased appetite, and feeling tired. For each item, respondents select the option that best describes how they felt over the previous 2 weeks. Every question has anchors arranged according to severity, and the score ranges from 0 to 3 points. The higher the total score is, the more severe the depression symptoms are. A total score of 0-13 points is in the normal range, 14-19 implies mild depression, 20-28 moderate depression, and 29-63 severe depression.